CLINICAL TRIAL: NCT04209816
Title: Genetic Regulation of Lipid Pathways Contributing to Non-alcoholic Fatty Liver and Atherogenic Dyslipidemia
Brief Title: Genetic Pathways Leading to Fatty Liver and Atherogenic Dyslipidemia
Acronym: VARKIN
Status: Enrolling by invitation | Type: Observational
Sponsor: Marja-Riitta Taskinen (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Marja-Riitta Taskinen, Professor, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Other Study IDs: HUS/53/2017
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Non-alcoholic Fatty Liver; Atherogenic Dyslipidemia; Insulin Resistance
Keywords: Non-alcoholic Fatty Liver; Apoproteins; Genetic variants
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- ApoC-III LOF: Carriers of apo-CIII loss-of-function mutation
  Interventions: Diagnostic Test: Lipoprotein kinetics
- ApoC-III GOF: Carriers of apo-CIII gain-of-function mutation
  Interventions: Diagnostic Test: Lipoprotein kinetics
- TM6SF2-KK: Carriers of TM6SF2 E167K mutation
  Interventions: Diagnostic Test: Lipoprotein kinetics
- PNLPLA3-MM: Carriers of PNLPLA3 I148M mutation
  Interventions: Diagnostic Test: Lipoprotein kinetics
- Control: No ApoC-III, TM6SF2 E167K or PNLPLA3 I148M mutation
  Interventions: Diagnostic Test: Lipoprotein kinetics
- ApoE variants: Carriers of E2/2, E3/3 or E4/4 mutation
  Interventions: Diagnostic Test: Lipoprotein kinetics
- LIPG: LIPG gene LOF or GOF variant carriers
  Interventions: Diagnostic Test: Lipoprotein kinetics
- ANGPTL3 or ANGPTL8: ANGPTL3 and ANGPTL8 gene LOF or GOF variant carriers

INTERVENTIONS:
Diagnostic Test: Lipoprotein kinetics — Lipoprotein kinetic apply protocol that endogenously label proteins and fatty acids with stable isotope-labeled amino acid and glycerol tracers. De novo lipogenesis is measured after ingestion of deuterated water to measure newly formed fatty acids in VLDL. Liver fat is measured with magnetic resonance spectroscopy and lipolytic enzymes with heparin test.
  Other Names: Measurement of de novo lipogenesis; Measurement of lipolytic activity; Measurement of liver fat
  Groups: ApoC-III GOF; ApoC-III LOF; ApoE variants; Control; LIPG; PNLPLA3-MM; TM6SF2-KK

SUMMARY:
The aims of the study are:

1. To investigate if carriers of apolipoprotein (apo) CIII loss-of-function (LOF) mutations produce less apo-CIII that results in reduction of large very low-density lipoprotein (VLDL) particle secretion as compared to non-carriers of these variants and compare the results with carriers of apo-CIII gain-of-function (GOF) to elucidate the role of apo-CIII in hepatic lipid metabolism.
2. To study if carriers of the TM6SF2 E167K and PNLPLA3 I148M mutations produce less large VLDL particles to transport fat out of the liver as compared to non-carriers.
3. To test whether the specific mutations in the apo-CIII, TM6SF2 and PNLPLA3 genes are reflected in changes of liver de novo lipogenesis (DNL), liver fat, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), plasma lipid and apolipoprotein kinetics and fasting concentrations in carriers of the TM6SF2 E167K and PNLPLA3 I148M mutations as compared to non-carriers.
4. To study the effects of APOE, angiopoietin (ANGPTL3 and ANGPTL8) or endothelial lipase (LIPG) genotypes on liver fat metabolism, lipid and apolipoprotein metabolism and lipid phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided written consent
* apo-CIII loss-of-function mutation (heterozygous) or apo-CIII gain-of-function mutations (heterozygous) or TM6SF2 E167K mutation (homozygous) or PNLPLA3 I148M or apoE or LIPG or ANGPTL3 or ANGPTL8 LOF and GOF variants. Control group without any of known risk variants in these genes.
* Hemoglobin A1c < 6.5%
* Body mass index between 18.5 and 40 kg/m²
* Estimated glomerular filtration rate > 60 ml/min/1.73 m² at inclusion

Exclusion Criteria:

* Patients with Type 1 and 2 diabetes, BMI > 40 kg/m2,
* ApoE2/2 phenotype, thyrotropin concentration outside normal range,
* Lipid-lowering drugs
* Blood pressure >160 mmHg systolic and/or > 105 diastolic mmHg
* Liver failure or abnormal liver function tests >3 x upper limit of normal
* Intestinal disease
* Pregnancy, breastfeeding
* Patients with volume depletion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory outpatients who are recruited from our previous study investigating familial dyslipidemia where exome sequency has been performed to explore genes involved in lipid metabolism (HUCH Ethics Committee, Department of Medicine: 108/1996, follow-up studies Dnro 170/E5/02, Drno 215/13/03/01/2009, Drno 144/13/03/01/2011 and HUCH Coordinating Ethics Committee Drno 184/13/03/00/2012, and Drno 183/13/03/00/2012). All subjects who have given oral consent that they can be informed about new studies focused on lipid metabolism will be contacted. To recruite the subjects we will use the invitation letter and follow up all the policy as stipulated in the Finnish biobank law (688/2012) (http//nationalbiobanks.fi/index.php./studies2/7-finrisk).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Difference in the rate of production of VLDL Apo B | Baseline
  Production rate, mg/day
Difference in the rate of production of VLDL Triglycerides | Baseline
  Production rate, mg/kg/day
Difference in the rate of production of VLDL ApoC-III and apoE | Baseline
  Production rate, mg/kg/day
Difference in the Fractional Catabolic Rate of VLDL Apo B | Baseline
  Rate of disappearance, pools/day
Difference in the Fractional Catabolic Rate of VLDL Triglycerides | Baseline
  Rate of disappearance, pools/day
Difference in the Fractional Catabolic Rate of VLDL ApoC-III and apoE | Baseline
  Rate of disappearance, pools/day
Difference in de novo lipogenesis | Baseline
  Measure of newly synthesized triglycerides in VLDL, μmol/l
Difference in liver fat | Baseline
  Percentage of liver fat measured with magnetic resonance spectroscopy
Difference in atherogenic dyslipidemia | Baseline
  Remnant lipoproteins and lipoprotein fraction composition, mg/L
Difference in insulin resistance | Baseline
  Calculated Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Difference in apoprotein A concentration | Baseline
  ApoA, mg/dl
Difference in apoprotein B concentration | Baseline
  ApoB, mg/dl
Difference in apoprotein C concentration | Baseline
  ApoC, mg/dl
Difference in apoprotein E concentration | Baseline
  ApoE, mg/dl
Difference in the rate of production and Fractional Catabolic Rate of intermediate-density Apo B | Baseline
  Rate of turnover, pools/day
Difference in the rate of production and Fractional Catabolic Rate of low-density lipoprotein Apo B | Baseline
  Rate of turnover, pools/day
Lipolytic activity | Baseline
  Measured lipoprotein lipase activity, mU/ml
Hepatic lipase activity | Baseline
  Measured hepatic lipase activity, mU/ml

CONTACTS AND LOCATIONS:
Locations (2):
- RPU Clinical and Molecular Metabolism, Biomedicum, Helsinki, Finland
- Wallenberg Laboratory, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taskinen MR, Bjornson E, Matikainen N, Soderlund S, Ramo J, Ainola MM, Hakkarainen A, Sihlbom C, Thorsell A, Andersson L, Bergh PO, Henricsson M, Romeo S, Adiels M, Ripatti S, Laakso M, Packard CJ, Boren J. Postprandial metabolism of apolipoproteins B48, B100, C-III, and E in humans with APOC3 loss-of-function mutations. JCI Insight. 2022 Oct 10;7(19):e160607. doi: 10.1172/jci.insight.160607. PMID 36040803